CLINICAL TRIAL: NCT00389493
Title: Maximizing Treatment Outcome in OCD
Brief Title: Risperidone or Cognitive-Behavioral Therapy for Improving Medication Treatment for Obsessive-compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #5188/#6258R; R01MH045436-02 (NIH); DSIR 83-ATAS; R01MH045436 (NIH); R01MH045404 (NIH)
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Results first posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2013-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; Augmentation; Antipsychotics; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Participants will receive treatment with risperidone
  Interventions: Drug: Risperidone
- 2 (Active Comparator): Participants will receive exposure and ritual prevention therapy (EX/RP)
  Interventions: Behavioral: Exposure/ritual prevention therapy (EX/RP)
- 3 (Placebo Comparator): Participants will receive treatment with the placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — Dosage of 0.5 mg to 4.0 mg per day as tolerated
  Other Names: Risperdal
  Arms: 1
Behavioral: Exposure/ritual prevention therapy (EX/RP) — EX/RP is a form of cognitive behavioral therapy. Participants assigned to EX/RP will attend therapy sessions twice per week. In EX/RP, participants will be exposed to feared objects or ideas, and will be encouraged not to carry out a compulsive response.
  Other Names: EX/RP
  Arms: 2
Drug: Placebo — Placebo capsules will be identical in appearance to those of risperidone.
  Other Names: PBO
  Arms: 3

SUMMARY:
This study will compare the short- and long-term effectiveness of two common therapies in improving serotonin reuptake inhibitor treatment in people with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a common psychiatric illness. People with OCD experience unwelcome thoughts, known as obsessions, and feel compelled to perform repetitive behaviors, or compulsions. Impairment due to OCD symptoms ranges from mild to severe, and sometimes can be disabling. The only medications proven effective for OCD are serotonin reuptake inhibitors (SRIs), but even with SRI treatment, most patients continue to experience significant OCD symptoms, impaired functioning, and diminished quality of life. Cognitive-behavioral therapy (CBT), a talking therapy that focuses on altering a person's thoughts and behaviors, and the medication risperidone have both been commonly used for augmenting SRI treatment for OCD. This study will compare the short- and long-term effectiveness of exposure and ritual prevention (EX/RP), a type of CBT, and risperidone in augmenting SRI treatment in people with OCD.

Participants in this double-blind study will be randomly assigned to receive EX/RP, risperidone, or placebo in conjunction with their regular SRI medication. All participants will remain on their regular SRI at a stable dose. During the first 2 months of the study, participants assigned to EX/RP will attend therapy sessions twice per week. In EX/RP, participants will be exposed to feared objects or ideas, and will be encouraged not to carry out a compulsive response. Participants assigned to risperidone or placebo will meet with a psychiatrist once every 1 to 2 weeks. At the end of 8 weeks, all participants' OCD symptom severity will be assessed. During this time, participants who have responded to treatment will continue receiving the same treatment for an additional 24 weeks. Participants assigned to EX/RP will meet with a therapist no more than 15 times total, and participants receiving risperidone or placebo will meet with a psychiatrist once every 4 weeks. Outcomes will be reassessed at study completion.

Ortho McNeil Janssen Scientific Affairs, LLC are providing medication and placebos for this study.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00045903

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of OCD
* Currently on a stable and adequate dose of an SRI
* Sufficient severity of symptoms to warrant additional augmentation treatment

Exclusion Criteria:

* Medical or psychiatric conditions that would make participation in the study unsafe
* Currently receiving psychotherapy elsewhere at the time of study entry
* Previously (within 12 weeks prior to study entry) attended 8 or more sessions of EX/RP within a 2-month period or received at least 4 weeks of antipsychotic augmentation while on an adequate SRI dose
* Currently being treated with an SRI for the first time and has not yet responded, but has not tried another SRI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blair Simpson, MD, PhD, Principal Investigator — New York State Psychiatric Institute; Edna Foa, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - New York State Psychiatric Institute, New York, New York
  - University of Pennsylvania Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Simpson HB, Foa EB, Liebowitz MR, Huppert JD, Cahill S, Maher MJ, McLean CP, Bender J Jr, Marcus SM, Williams MT, Weaver J, Vermes D, Van Meter PE, Rodriguez CI, Powers M, Pinto A, Imms P, Hahn CG, Campeas R. Cognitive-behavioral therapy vs risperidone for augmenting serotonin reuptake inhibitors in obsessive-compulsive disorder: a randomized clinical trial. JAMA Psychiatry. 2013 Nov;70(11):1190-9. doi: 10.1001/jamapsychiatry.2013.1932. PMID 24026523
- [Derived] McLean CP, Zandberg LJ, Van Meter PE, Carpenter JK, Simpson HB, Foa EB. Exposure and response prevention helps adults with obsessive-compulsive disorder who do not respond to pharmacological augmentation strategies. J Clin Psychiatry. 2015 Dec;76(12):1653-7. doi: 10.4088/JCP.14m09513. PMID 26613263
- [Derived] Foa EB, Simpson HB, Rosenfield D, Liebowitz MR, Cahill SP, Huppert JD, Bender J Jr, McLean CP, Maher MJ, Campeas R, Hahn CG, Imms P, Pinto A, Powers MB, Rodriguez CI, Van Meter PE, Vermes D, Williams MT. Six-month outcomes from a randomized trial augmenting serotonin reuptake inhibitors with exposure and response prevention or risperidone in adults with obsessive-compulsive disorder. J Clin Psychiatry. 2015 Apr;76(4):440-6. doi: 10.4088/JCP.14m09044. PMID 25375780
- [Derived] Farris SG, McLean CP, Van Meter PE, Simpson HB, Foa EB. Treatment response, symptom remission, and wellness in obsessive-compulsive disorder. J Clin Psychiatry. 2013 Jul;74(7):685-90. doi: 10.4088/JCP.12m07789. PMID 23945445
- See also: Click here for the Columbia University Obsessive-Compulsive Disorder Research Clinic website — http://www.columbia-ocd.org/
- See also: Click here for the University of Pennsylvania Center for the Treatment and Study of Anxiety website — http://www.med.upenn.edu/ctsa/
- See also: Click here to view the ClinicalTrials.gov record of this trial's parent study — http://www.clinicaltrials.gov/show/NCT00045903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized clinical trial (conducted January 2007-August 2012) at 2 academic outpatient research clinics that specialize in OCD and anxiety disorders. Patients (aged 18-70 years) were eligible if they had OCD of at least moderate severity despite a therapeutic SRI dose for at least 12 weeks prior to entry.
Groups:
- Treatment With Risperidone: Participants will receive treatment with risperidone
  Risperidone : Dosage of 0.5 mg to 4.0 mg per day as tolerated
- Treatment With Exposure/Response Prevention: Participants will receive exposure and response prevention therapy
  Exposure/ritual prevention therapy (EX/RP) : EX/RP is a form of cognitive behavioral therapy. Participants assigned to EX/RP will attend therapy sessions twice per week. In EX/RP, participants will be exposed to feared objects or ideas, and will be encouraged not to carry out a compulsive response.
- Treatment With Pill Placebo: Participants will receive treatment with the placebo
  Placebo : Placebo capsules will be identical in appearance to those of risperidone.
Period: Overall Study
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Started | 40 | 40 | 20
Completed | 37 | 32 | 17
Not Completed | 3 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo | Total
Number analyzed (Participants) | 40 | 40 | 20 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 20 | 100
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (10.8) | 34.3 (12.7) | 33.4 (10.4) | 33.9 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 6 | 48
  Male | 19 | 19 | 14 | 52
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 20 | 100

OUTCOME MEASURES:

1. Primary Outcome: Score on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
Description: Y-BOCS ranges from 0-40, with 0 meaning no symptoms and higher numbers meaning greater symptom severity
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment With Risperidone: Participants received treatment with risperidone Risperidone : Dosage of 0.5 mg to 4.0 mg per day as tolerated Mean Y-BOCS score measured at week 8
- Treatment With Exposure/Response Prevention: Participants received exposure and response prevention therapy
  Exposure/ritual prevention therapy (EX/RP) : EX/RP is a form of cognitive behavioral therapy. Participants assigned to EX/RP will attend therapy sessions twice per week. In EX/RP, participants will be exposed to feared objects or ideas, and will be encouraged not to carry out a compulsive response.
  Mean Y-BOCS score measured at week 8
- Treatment With Pill Placebo: Participants received treatment with the placebo
  Placebo : Placebo capsules will be identical in appearance to those of risperidone.
  Mean Y-BOCS score measured at week 8
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Number analyzed (Participants) | 40 | 40 | 20
units on a scale
  Y-BOCS score at Week 0 | 26.1 (4.3) | 27.2 (3.9) | 25.9 (4.6)
  Y-BOCS score at Week 8 | 22.6 (8.8) | 13.0 (6.1) | 23.1 (6.9)

2. Secondary Outcome: Social Adjustment Scale-SR
Description: SAS-SR yields a mean score between 1 and 5; the higher the score, the more severe the social adjustment problems
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Number analyzed (Participants) | 40 | 40 | 20
units on a scale
  SAS-SR at Week 0 | 2.3 (0.4) | 2.3 (0.5) | 2.2 (0.7)
  SAS-SR at Week 8 | 2.2 (0.4) | 1.9 (0.4) | 2.1 (0.5)

3. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form
Description: QLESQ ranges from 14-70, with higher scores meaning more enjoyment and satisfaction with quality of life
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Number analyzed (Participants) | 40 | 40 | 20
units on a scale
  QLESQ-SF Week 0 | 52.3 (14.1) | 57.8 (16.2) | 56.1 (16.2)
  QLESQ-SF Week 8 | 55.1 (13.9) | 70.2 (14.2) | 62.6 (16.7)

4. Secondary Outcome: Hamilton Depression Rating Scale (Ham-D)
Description: Ham-D ranges from 0=no symptoms to 52 with higher numbers indicating more severe depression
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Number analyzed (Participants) | 40 | 40 | 20
units on a scale
  Ham-D at Week 0 | 9.8 (5.6) | 7.8 (6.1) | 7.7 (5.9)
  Ham-D at Week 8 | 8.0 (5.7) | 7.8 (6.1) | 7.7 (5.9)

5. Secondary Outcome: Brown Assessment of Beliefs (BABS)
Description: Scale ranges from 0 to 24 where 0 is "beliefs are false" and 24 is "convinced beliefs = reality"
Time Frame: Week 0 and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Number analyzed (Participants) | 40 | 40 | 20
units on a scale
  Week 0 | 5.7 (4.0) | 6.1 (4.6) | 5.3 (3.8)
  Week 8 | 4.5 (4.2) | 2.4 (2.9) | 4.3 (3.3)

ADVERSE EVENTS:
Arm/Group | Treatment With Risperidone | Treatment With Exposure/Response Prevention | Treatment With Pill Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 30/40 | 22/40 | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Risperidone (N=40) | Treatment With Exposure/Response Prevention (N=40) | Treatment With Pill Placebo (N=20)
Headache (Nervous system disorders) | 7 | 9 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2
Nausea (Gastrointestinal disorders) | 0 | 3 | 2
Sweating (General disorders) | 1 | 4 | 3
Photophobia (Eye disorders) | 5 | 3 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 2
Lightheadedness (Nervous system disorders) | 5 | 6 | 2
Dry Mouth (Gastrointestinal disorders) | 10 | 2 | 5
Blurry Vision (Eye disorders) | 5 | 1 | 2
Decreased Libido (Reproductive system and breast disorders) | 9 | 6 | 1
Anorgasmia/Erectile Failure (Reproductive system and breast disorders) | 6 | 4 | 0
Impaired Coordination (Nervous system disorders) | 1 | 1 | 2
Fatigue (Nervous system disorders) | 9 | 8 | 4
Nervousness (Nervous system disorders) | 8 | 6 | 4
Insomnia (Nervous system disorders) | 7 | 5 | 3
Tremor (Nervous system disorders) | 0 | 3 | 3
Weight Gain (Gastrointestinal disorders) | 13 | 7 | 2
Weight Loss (Gastrointestinal disorders) | 3 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Urinary Dysfunction (Renal and urinary disorders) | 3 | 1 | 1
Changes in breasts (Reproductive system and breast disorders) | 3 | 0 | 0
Increased thirst (Gastrointestinal disorders) | 6 | 1 | 4
Somnolence (Nervous system disorders) | 7 | 7 | 4
Extrapyramidal symptoms (Nervous system disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes